CLINICAL TRIAL: NCT00755014
Title: Taipei Veterans General Hospital
Brief Title: Study Effect of Red Wine Consumption on Endothelial Progenitor Cells and Endothelial Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Medial Resource and Education, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHIRB No: 96-01-11A
Record Dates: First submitted 2008-09-15; First posted 2008-09-18 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Endothelial Progenitor Cells Numbers; Endothelial Function (FMD)
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Experimental): Forty subjects are randomized to a group (n=20) that consumed red wine (100 ml) or a group (n=20) that consumed beer (250 ml) daily for 3 weeks
  Interventions: Other: red wine

INTERVENTIONS:
Other: red wine — One group (n=20) that consumed red wine (100 ml) daily for 3 weeks Another group (n=20) that consumed beer (250 ml) daily for 3 weeks
  Other Names: The red wine used is "Vin De Pays D'OC" (12.5% ethanol), a cabernet sauvignon from France; The beer used was Taiwan Beer (5% alcohol) from Taiwan.

SUMMARY:
Light-to-moderate alcohol consumption has been associated with a reduction of cardiovascular events, and red wine seems to offer more benefits than any other type of alcoholic beverages. However, the relationship between red wine consumption and endothelial progenitor cells (EPCs) remains unclear. The investigators examine whether intake of red wine could enhance the number or functional capacity of circulating EPCs by upregulation of nitric oxide (NO) bioavailability.

DETAILED DESCRIPTION:
Moderate ethanol intake from any type of beverage has been shown to improve lipoprotein metabolism and lower cardiovascular mortality risk, but red wine, with its abundant antioxidant contents, seems to confer additional healthy benefits. Previous studies indicated that the beneficial effects of red wine are derived from increased endothelium-derived nitric oxide (NO), implying that enhanced NO bioavailability may mediate the cardiovascular protection provided by red wine.

Increasing evidence suggests that the injured endothelial monolayer is regenerated partly by circulating bone marrow derived-endothelial progenitor cells (EPCs), which accelerate reendothelialization and protect against the initiation and progression of atherosclerosis. Clinical studies demonstrated that the number of circulating EPCs predicts the occurrence of cardiovascular events and death from cardiovascular causes and may help to identify patients at increased cardiovascular risk. Although many epidemiologic studies have indicated that light-to-moderate consumption of red wine can reduce the incidence of CAD, the multifarious effects of red wine on circulating EPCs and endothelial function remain to be determined. Therefore, we design this study to test the hypothesis that intake of red wine can enhance the number and functional capacity of EPCs through increasing NO bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* Forty young healthy subjects with no cardiovascular risk factors

Exclusion Criteria:

* History of hypertension
* Diabetes mellitus
* Symptoms of CAD
* Smoking
* Chronic renal insufficiency (serum creatinine > 1.5 mg/dl)
* Inflammatory or liver diseases
* Regular alcohol consumption (drinking more than 20 g of ethanol per week)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Number of endothelial progenitor cells, endothelial function (FMD) | VGH-97DHA0100127

SECONDARY OUTCOMES:
Plasma NO, hsCRP, ADMA, TNF-a, adiponectin, ox-LDL levels | VGH-97DHA0100127

CONTACTS AND LOCATIONS:
Overall Officials: Shing-Jong Lin, MD, PhD, Principal Investigator — Division of Cardiology, Taipei Veterans General Hospital; Po-Hsun Huang, MD, Study Director — Division of Cardiology, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans Generla Hospital, Taipei, Taiwan